CLINICAL TRIAL: NCT04410406
Title: A Clinical Trial to Assess the Safety and Efficacy of Moxidectin Combination Treatments vs. Ivermectin Combination Treatments for Bancroftian Filariasis
Brief Title: Moxidectin for LF, Cote d'Ivoire (DOLF)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Washington University School of Medicine (Other)
Collaborators: Case Western Reserve University (Other); Centre Suisse de Recherches Scientifiques en Cote d'Ivoire (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 202005076
Record Dates: First submitted 2020-05-27; First posted 2020-06-01 (Actual); Results first posted 2026-01-29 (Actual); Last update posted 2026-01-29 (Actual); Status verified 2026-01

CONDITIONS: Lymphatic Filariasis
Keywords: moxidectin; ivermectin
MeSH Terms: conditions — Elephantiasis, Filarial | interventions — Ivermectin; Diethylcarbamazine; Albendazole; moxidectin

STUDY DESIGN:
Intervention Model Description: This trial is a single-site, Phase III, randomized, open-label, masked-observer superiority trial with four treatment arms (IA, MoxA, IDA, and MoxDA). Block randomization by gender will be used to assign treatment arms.
Masking Description: Recognizing that number and appearance of tablets received in each study arm will be noticeably different, this study will not be completely masked to participants or care providers. To minimize bias, administration of study medications will be performed by a staff member with no role in assessing AEs. AE assessments and all other outcome measures will be assessed by observers masked to the treatment assignment as best as possible.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (4):
- IA (Ivermectin + Albendazole) (Active Comparator): Participants will receive one oral dose of Ivermectin (IVM) 200 µg/kg + Albendazole (ABZ) 400 mg (IA) annually for 24 months.
  Interventions: Drug: Ivermectin; Drug: Albendazole
- MoxA (Moxidectin + Albendazole) (Active Comparator): Participants will receive one oral dose of Mox 8 mg + ABZ 400 mg. Participants who are Mf positive at 24 months will be retreated with MoxA at the same dosage.
  Interventions: Drug: Albendazole; Drug: Moxidectin
- IDA (Ivermectin + Diethylcarbamazine + Albendazole) (Active Comparator): Participants will receive one oral dose of IVM 200 µg/kg + Diethylcarbamazine (DEC) 6mg/kg + ABZ 400 mg. Participants who are Mf positive at 24 months will be retreated with IDA at the same dosage.
  Interventions: Drug: Ivermectin; Drug: Diethylcarbamazine; Drug: Albendazole
- MoxDA (Moxidectin + Diethylcarbamazine + Albendazole) (Active Comparator): Participants will receive one oral dose of Mox 8 mg + DEC 6mg/kg + ABZ 400 mg. Participants who are Mf positive at 24 months will be retreated with MoxDA at the same dosage.
  Interventions: Drug: Diethylcarbamazine; Drug: Albendazole; Drug: Moxidectin

INTERVENTIONS:
Drug: Ivermectin — Ivermectin (IVM) 200 µg/kg
  Other Names: Stromectol
  Arms: IA (Ivermectin + Albendazole); IDA (Ivermectin + Diethylcarbamazine + Albendazole)
Drug: Diethylcarbamazine — Diethylcarbamazine (DEC) 6mg/kg
  Other Names: Diethylcarbamazine citrate; Hetrazan
  Arms: IDA (Ivermectin + Diethylcarbamazine + Albendazole); MoxDA (Moxidectin + Diethylcarbamazine + Albendazole)
Drug: Albendazole — Albendazole (ABZ) 400 mg
Drug: Moxidectin — Moxidectin (Mox) 8 mg
  Arms: MoxA (Moxidectin + Albendazole); MoxDA (Moxidectin + Diethylcarbamazine + Albendazole)

SUMMARY:
The purpose of this study is to determine whether moxidectin (Mox) will be more effective than ivermectin (IVM) when used in single-dose combination therapies for lymphatic filariasis (LF).

DETAILED DESCRIPTION:
This study will test the hypothesis that Moxidectin combination therapies are superior to ivermectin combination therapies for achieving sustained clearance of W. bancrofti microfilaremia.

This trial is designed as single-site, Phase III, randomized, open-label, masked-observer superiority trial with four treatment arms: ivermectin + albendazole (IA), moxidectin + albendazole (MoxA), ivermectin + diethylcarbamazine + albendazole (IDA), and moxidectin + diethylcarbamazine + albendazole (MoxDA). The primary endpoint is the proportion of participants achieving complete clearance of microfilaremia at 12 months (IA vs. MoxA comparison) or 24 months (IDA vs. MoxDA comparison). Block randomization by gender will be used to assign treatment arms.

The first 48 participants (12 each arm) will be treated at Agboville Hospital in Cote d'Ivoire at the Centre de Recherche de Filariose with inpatient AE monitoring and collection of post-treatment plasma drug levels (Part 1). For Part 1, active AE surveillance will be conducted in the hospital on days 1, 2, and 3, post-treatment, and in the participant's village of residence on day 7 post-treatment and passive surveillance will be conducted by trained village health workers on days 4-6. An interim safety analysis will take place after Part 1. If no safety concerns are identified, the remainder of the participants will be treated in their home villages, with active AE monitoring on days 1 and 2 post-treatment (Part 2) with passive surveillance by trained village health workers on days 3-7. Any participant in either Part 1 or Part 2 experiencing AEs of grade 2 or higher will be followed until adverse event (AE) severity falls below grade 2. Follow-up assessments for efficacy of treatments for all participants (Parts 1 and 2) will be conducted at 6, 12, 24, and 36 months.

The study includes both safety and efficacy analyses. The safety assessment (Part 1 only) ends 7 days after treatment (unless AEs remain grade 2 or higher). The efficacy assessment (Parts 1 and 2 combined) ends when participants are retested for filarial infection 36 months post-treatment. Participants in the IA arm will receive IA annually (standard of care). Participants in the other arms will receive the assigned treatment at baseline; those found to be microfilaremic at 24 months post-treatment will be retreated with the same treatment received at baseline. If clearance of microfilariae (Mf) at 12 months in the IA arm is superior to Mf clearance in the MoxA arm, the MoxA group will be switched to annual IA treatment.

The study design does not currently include stratification, nor do any sub-studies. However, the study may stratify based on pre-treatment Mf levels if high variability among pre-screening Mf counts is observed.

ELIGIBILITY:
Inclusion Criteria:

* Provision of signed and dated informed consent form
* Male or female, aged 18-70 years
* In good general health as evidenced by medical history
* Peripheral night blood W. bancrofti Mf levels ≥40 Mf/mL
* No history of taking antifilarial medications in past 12 months
* Resident of the study area with no plans to change residence in the next 36 months
* For women of childbearing potential, willing to use appropriate method of contraception for one month following each treatment

Exclusion Criteria:

* Pregnancy or currently breastfeeding
* Known allergic reactions to any of the study medications
* Evidence of severe or systemic comorbidities (aside from features of filarial disease), as judged by the principal investigator
* Baseline biochemical abnormalities, as indicated by AST, ALT, or creatinine > 2 times the upper limit of normal
* Evidence of urinary tract infection as indicated by 3+ nitrites on dipstick (individuals with 1+ or 2+ nitrites will not be excluded) or underlying chronic kidney disease as indicated by 3+ protein or 3+ blood on urine dipstick exam
* Hgb < 7 gm/dL (any such individuals will be referred to the local health center for evaluation and treatment)
* Positive skin snip for onchocerciasis

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 164 (Actual)
Dates: Start 2020-08-20 (Actual); Primary Completion 2024-10-01 (Actual); Study Completion 2024-10-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Philip Budge, MD, PhD, Principal Investigator — Washington University School of Medicine; Catherine Bjerum, MD, MPH, Principal Investigator — Case Western Reserve University; Toki Pascal Gabo, MD, Principal Investigator — Regional Hospital of Agboville, Southern Cote d'Ivoire; Benjamin Koudou, PhD, Principal Investigator — Regional Hospital of Agboville, Southern Cote d'Ivoire
Locations (1):
- Regional Hospital of Agboville, Southern Cote d'Ivoire, Agboville, Côte d’Ivoire

IPD SHARING:
Plan to Share IPD: Yes
De-identified datasets used for published results will be shared publically through a journal or other open source data repository so that the broader scientific community can access it. Datasets used for published results will be shared publically through a journal or other open source data repository so that the broader scientific community can access it. Only de-identified data will be shared outside of the study team.

REFERENCES:
- [Background] Opoku NO, Bakajika DK, Kanza EM, Howard H, Mambandu GL, Nyathirombo A, Nigo MM, Kasonia K, Masembe SL, Mumbere M, Kataliko K, Larbelee JP, Kpawor M, Bolay KM, Bolay F, Asare S, Attah SK, Olipoh G, Vaillant M, Halleux CM, Kuesel AC. Single dose moxidectin versus ivermectin for Onchocerca volvulus infection in Ghana, Liberia, and the Democratic Republic of the Congo: a randomised, controlled, double-blind phase 3 trial. Lancet. 2018 Oct 6;392(10154):1207-1216. doi: 10.1016/S0140-6736(17)32844-1. Epub 2018 Jan 18. PMID 29361335
- [Background] Ichimori K, King JD, Engels D, Yajima A, Mikhailov A, Lammie P, Ottesen EA. Global programme to eliminate lymphatic filariasis: the processes underlying programme success. PLoS Negl Trop Dis. 2014 Dec 11;8(12):e3328. doi: 10.1371/journal.pntd.0003328. eCollection 2014 Dec. No abstract available. PMID 25502758
- [Background] Ottesen EA, Duke BO, Karam M, Behbehani K. Strategies and tools for the control/elimination of lymphatic filariasis. Bull World Health Organ. 1997;75(6):491-503. PMID 9509621
- [Background] Ottesen EA. Lymphatic filariasis: Treatment, control and elimination. Adv Parasitol. 2006;61:395-441. doi: 10.1016/S0065-308X(05)61010-X. PMID 16735170
- [Background] Thomsen EK, Sanuku N, Baea M, Satofan S, Maki E, Lombore B, Schmidt MS, Siba PM, Weil GJ, Kazura JW, Fleckenstein LL, King CL. Efficacy, Safety, and Pharmacokinetics of Coadministered Diethylcarbamazine, Albendazole, and Ivermectin for Treatment of Bancroftian Filariasis. Clin Infect Dis. 2016 Feb 1;62(3):334-341. doi: 10.1093/cid/civ882. Epub 2015 Oct 20. PMID 26486704
- [Background] King CL, Suamani J, Sanuku N, Cheng YC, Satofan S, Mancuso B, Goss CW, Robinson LJ, Siba PM, Weil GJ, Kazura JW. A Trial of a Triple-Drug Treatment for Lymphatic Filariasis. N Engl J Med. 2018 Nov 8;379(19):1801-1810. doi: 10.1056/NEJMoa1706854. PMID 30403937
- [Background] Edi C, Bjerum CM, Ouattara AF, Chhonker YS, Penali LK, Meite A, Koudou BG, Weil GJ, King CL, Murry DJ. Pharmacokinetics, safety, and efficacy of a single co-administered dose of diethylcarbamazine, albendazole and ivermectin in adults with and without Wuchereria bancrofti infection in Cote d'Ivoire. PLoS Negl Trop Dis. 2019 May 20;13(5):e0007325. doi: 10.1371/journal.pntd.0007325. eCollection 2019 May. PMID 31107869
- [Background] Irvine MA, Stolk WA, Smith ME, Subramanian S, Singh BK, Weil GJ, Michael E, Hollingsworth TD. Effectiveness of a triple-drug regimen for global elimination of lymphatic filariasis: a modelling study. Lancet Infect Dis. 2017 Apr;17(4):451-458. doi: 10.1016/S1473-3099(16)30467-4. Epub 2016 Dec 22. PMID 28012943
- [Background] Kyelem D, Biswas G, Bockarie MJ, Bradley MH, El-Setouhy M, Fischer PU, Henderson RH, Kazura JW, Lammie PJ, Njenga SM, Ottesen EA, Ramaiah KD, Richards FO, Weil GJ, Williams SA. Determinants of success in national programs to eliminate lymphatic filariasis: a perspective identifying essential elements and research needs. Am J Trop Med Hyg. 2008 Oct;79(4):480-4. PMID 18840733
- [Background] Molyneux DH, Hopkins A, Bradley MH, Kelly-Hope LA. Multidimensional complexities of filariasis control in an era of large-scale mass drug administration programmes: a can of worms. Parasit Vectors. 2014 Aug 15;7:363. doi: 10.1186/1756-3305-7-363. PMID 25128408
- [Background] Horton J. Albendazole: a broad spectrum anthelminthic for treatment of individuals and populations. Curr Opin Infect Dis. 2002 Dec;15(6):599-608. doi: 10.1097/00001432-200212000-00008. PMID 12821837
- [Background] Horton J, Witt C, Ottesen EA, Lazdins JK, Addiss DG, Awadzi K, Beach MJ, Belizario VY, Dunyo SK, Espinel M, Gyapong JO, Hossain M, Ismail MM, Jayakody RL, Lammie PJ, Makunde W, Richard-Lenoble D, Selve B, Shenoy RK, Simonsen PE, Wamae CN, Weerasooriya MV. An analysis of the safety of the single dose, two drug regimens used in programmes to eliminate lymphatic filariasis. Parasitology. 2000;121 Suppl:S147-60. doi: 10.1017/s0031182000007423. PMID 11386686
- [Background] Kitzman D, Cheng KJ, Fleckenstein L. HPLC assay for albendazole and metabolites in human plasma for clinical pharmacokinetic studies. J Pharm Biomed Anal. 2002 Oct 15;30(3):801-13. doi: 10.1016/s0731-7085(02)00382-5. PMID 12367706
- [Background] Geary TG. Ivermectin 20 years on: maturation of a wonder drug. Trends Parasitol. 2005 Nov;21(11):530-2. doi: 10.1016/j.pt.2005.08.014. Epub 2005 Aug 26. PMID 16126457
- [Background] Moreno Y, Nabhan JF, Solomon J, Mackenzie CD, Geary TG. Ivermectin disrupts the function of the excretory-secretory apparatus in microfilariae of Brugia malayi. Proc Natl Acad Sci U S A. 2010 Nov 16;107(46):20120-5. doi: 10.1073/pnas.1011983107. Epub 2010 Nov 1. PMID 21041637
- [Background] Awadzi K, Edwards G, Opoku NO, Ardrey AE, Favager S, Addy ET, Attah SK, Yamuah LK, Quartey BT. The safety, tolerability and pharmacokinetics of levamisole alone, levamisole plus ivermectin, and levamisole plus albendazole, and their efficacy against Onchocerca volvulus. Ann Trop Med Parasitol. 2004 Sep;98(6):595-614. doi: 10.1179/000349804225021370. PMID 15324466
- [Background] Kitzman D, Wei SY, Fleckenstein L. Liquid chromatographic assay of ivermectin in human plasma for application to clinical pharmacokinetic studies. J Pharm Biomed Anal. 2006 Mar 3;40(4):1013-20. doi: 10.1016/j.jpba.2005.08.026. Epub 2005 Oct 19. PMID 16242280
- [Background] Awadzi K, Edwards G, Duke BO, Opoku NO, Attah SK, Addy ET, Ardrey AE, Quartey BT. The co-administration of ivermectin and albendazole--safety, pharmacokinetics and efficacy against Onchocerca volvulus. Ann Trop Med Parasitol. 2003 Mar;97(2):165-78. doi: 10.1179/000349803235001697. PMID 12803872
- [Background] Bolla S, Boinpally RR, Poondru S, Devaraj R, Jasti BR. Pharmacokinetics of diethylcarbamazine after single oral dose at two different times of day in human subjects. J Clin Pharmacol. 2002 Mar;42(3):327-31. doi: 10.1177/00912700222011247. PMID 11865970
- [Background] Geary TG, Woo K, McCarthy JS, Mackenzie CD, Horton J, Prichard RK, de Silva NR, Olliaro PL, Lazdins-Helds JK, Engels DA, Bundy DA. Unresolved issues in anthelmintic pharmacology for helminthiases of humans. Int J Parasitol. 2010 Jan;40(1):1-13. doi: 10.1016/j.ijpara.2009.11.001. Epub 2009 Nov 20. PMID 19932111
- [Background] McGarry HF, Plant LD, Taylor MJ. Diethylcarbamazine activity against Brugia malayi microfilariae is dependent on inducible nitric-oxide synthase and the cyclooxygenase pathway. Filaria J. 2005 Jun 2;4:4. doi: 10.1186/1475-2883-4-4. PMID 15932636
- [Background] Weil GJ, Bogus J, Christian M, Dubray C, Djuardi Y, Fischer PU, Goss CW, Hardy M, Jambulingam P, King CL, Kuttiat VS, Krishnamoorthy K, Laman M, Lemoine JF, O'Brian KK, Robinson LJ, Samuela J, Schechtman KB, Sircar A, Srividya A, Steer AC, Supali T, Subramanian S; DOLF IDA Safety Study Group. The safety of double- and triple-drug community mass drug administration for lymphatic filariasis: A multicenter, open-label, cluster-randomized study. PLoS Med. 2019 Jun 24;16(6):e1002839. doi: 10.1371/journal.pmed.1002839. eCollection 2019 Jun. PMID 31233507
- [Background] Budge PJ, Herbert C, Andersen BJ, Weil GJ. Adverse events following single dose treatment of lymphatic filariasis: Observations from a review of the literature. PLoS Negl Trop Dis. 2018 May 16;12(5):e0006454. doi: 10.1371/journal.pntd.0006454. eCollection 2018 May. PMID 29768412
- [Background] Weil GJ, Lammie PJ, Richards FO Jr, Eberhard ML. Changes in circulating parasite antigen levels after treatment of bancroftian filariasis with diethylcarbamazine and ivermectin. J Infect Dis. 1991 Oct;164(4):814-6. doi: 10.1093/infdis/164.4.814. PMID 1894943
- [Background] Chhonker YS, Sleightholm RL, Murry DJ. Bioanalytical method development and validation of moxidectin in plasma by LC-MS/MS: Application to in vitro metabolism. Biomed Chromatogr. 2019 Feb;33(2):e4389. doi: 10.1002/bmc.4389. Epub 2018 Oct 30. PMID 30238696
- [Background] Hertz MI, Nana-Djeunga H, Kamgno J, Jelil Njouendou A, Chawa Chunda V, Wanji S, Rush A, Fischer PU, Weil GJ, Budge PJ. Identification and characterization of Loa loa antigens responsible for cross-reactivity with rapid diagnostic tests for lymphatic filariasis. PLoS Negl Trop Dis. 2018 Nov 16;12(11):e0006963. doi: 10.1371/journal.pntd.0006963. eCollection 2018 Nov. PMID 30444866
- [Derived] Koudou GB, Bjerum CM, Ouattara FA, Gabo TP, Goss CW, Lew D, Dje NN, King CL, Fischer PU, Weil GJ, Budge PJ. Moxidectin combination therapies for lymphatic filariasis: an open-label, observer-masked, randomised controlled trial. Lancet Infect Dis. 2025 Oct;25(10):1075-1083. doi: 10.1016/S1473-3099(25)00111-2. Epub 2025 May 6. PMID 40345209
- [Derived] Bjerum CM, Koudou BG, Ouattara AF, Lew D, Goss CW, Gabo PT, King CL, Fischer PU, Weil GJ, Budge PJ. Safety and tolerability of moxidectin and ivermectin combination treatments for lymphatic filariasis in Cote d'Ivoire: A randomized controlled superiority study. PLoS Negl Trop Dis. 2023 Sep 18;17(9):e0011633. doi: 10.1371/journal.pntd.0011633. eCollection 2023 Sep. PMID 37721964
- [Derived] Chhonker YS, Bjerum C, Bala V, Ouattara AF, Koudou BG, Gabo TP, Alshehri A, Meite A, Fischer PU, Weil GJ, King CL, Budge PJ, Murry DJ. Pharmacokinetics of Moxidectin combined with Albendazole or Albendazole plus Diethylcarbamazine for Bancroftian Filariasis. PLoS Negl Trop Dis. 2023 Aug 24;17(8):e0011567. doi: 10.1371/journal.pntd.0011567. eCollection 2023 Aug. PMID 37616301
- See also: First new treatment for river blindness approved by U.S. FDA in 20 years 2018 [cited 2018 June 27]. — https://tdr.who.int/newsroom/news/item/14-06-2018-first-new-treatment-for-river-blindness-approved-by-u-s-fda-in-20-years

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | IA (Ivermectin + Albendazole) | MoxA (Moxidectin + Albendazole) | IDA (Ivermectin + Diethylcarbamazine + Albendazole) | MoxDA (Moxidectin + Diethylcarbamazine + Albendazole)
Started (Part 1 refers to participants that were followed for intensive safety monitoring through 7 days, while Part 2 were followed intensively through 48 hours, and then outpatient through 7 days. Participants from both Part 1 and 2 were included in the safety and efficacy analysis) | 41 | 40 | 41 | 42
Completed | 25 | 16 | 22 | 23
Not Completed | 16 | 24 | 19 | 19

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | IA (Ivermectin + Albendazole) | MoxA (Moxidectin + Albendazole) | IDA (Ivermectin + Diethylcarbamazine + Albendazole) | MoxDA (Moxidectin + Diethylcarbamazine + Albendazole) | Total
Number analyzed (Participants) | 29 | 22 | 32 | 30 | 113
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 29 | 22 | 32 | 30 | 113
  >=65 years | 0 | 0 | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 34.6 (10.6) | 37.3 (10.2) | 38.3 (11.9) | 39.7 (11.8) | 37 (11.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 2 | 2 | 4 | 10
  Male | 27 | 20 | 30 | 26 | 103
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  Côte D'Ivoire | 29 | 22 | 32 | 30 | 113
Blood microfilaria count, median (IQR) [Median (Inter-Quartile Range); unit: Mf/mL] | 342 [147 to 595] | 134 [98 to 318] | 204.5 [94 to 510.5] | 191.5 [83 to 312] | 209 [98 to 408]

OUTCOME MEASURES:

1. Primary Outcome: Clearance of Microfilaremia (IA vs. MoxA)
Description: The proportion of participants in IA and MoxA study arms with complete clearance of W. bancrofti microfilaremia at 12 months after treatment.
Time Frame: 12 months
Measure: Count of Participants; unit: Participants
Arm/Group | IA (Ivermectin + Albendazole) | MoxA (Moxidectin + Albendazole) | IDA (Ivermectin + Diethylcarbamazine + Albendazole) | MoxDA (Moxidectin + Diethylcarbamazine + Albendazole)
Number analyzed (Participants) | 25 | 19 | 28 | 28
Participants | 8 | 18 | 24 | 27

2. Primary Outcome: Clearance of Microfilaremia (IDA vs. MoxDA)
Description: The proportion of participants in IDA and MoxDA study arms with complete clearance of W. bancrofti microfilaremia at 24 months after treatment.
Time Frame: 24 months
Measure: Count of Participants; unit: Participants
Arm/Group | IA (Ivermectin + Albendazole) | MoxA (Moxidectin + Albendazole) | IDA (Ivermectin + Diethylcarbamazine + Albendazole) | MoxDA (Moxidectin + Diethylcarbamazine + Albendazole)
Number analyzed (Participants) | 25 | 16 | 22 | 23
Participants | 13 | 14 | 20 | 21

3. Secondary Outcome: Clearance of Microfilaremia
Description: The proportion of participants in each study arm with complete clearance of W. bancrofti microfilaremia at 6, 12, 24, & 36 months after treatment.
Time Frame: 6, 12, 24, & 36 months
Population: The number of participants analyzed at different time points differs because we were unable to follow everyone consistently in the field at all timepoints. In many cases, our participants may need to leave for farming or other seasonal obligations.
Measure: Count of Participants; unit: Participants
Arm/Group | IA (Ivermectin + Albendazole) | MoxA (Moxidectin + Albendazole) | IDA (Ivermectin + Diethylcarbamazine + Albendazole) | MoxDA (Moxidectin + Diethylcarbamazine + Albendazole)
Number analyzed (Participants) | 28 | 23 | 31 | 34
Participants
  6 months: number analyzed (Participants) | 28 | 18 | 27 | 34
  6 months | 8 | 15 | 20 | 24
  12 months: number analyzed (Participants) | 28 | 19 | 31 | 34
  12 months | 8 | 18 | 24 | 27
  24 months: number analyzed (Participants) | 25 | 16 | 22 | 23
  24 months | 13 | 14 | 20 | 21
  36 months | 22 | 20 | 30 | 32

4. Secondary Outcome: Change in Mf Counts
Description: Change in microfilariae counts (relative to baseline) at12 & 24 months
Time Frame: Assessed at Baseline, 6, 12, & 24 months; Reported at 12 and 24 months
Population: Mean microfilaria counts
Measure: Mean (95% Confidence Interval); unit: Mf/mL
Arm/Group | IA (Ivermectin + Albendazole) | MoxA (Moxidectin + Albendazole) | IDA (Ivermectin + Diethylcarbamazine + Albendazole) | MoxDA (Moxidectin + Diethylcarbamazine + Albendazole)
Number analyzed (Participants) | 25 | 19 | 28 | 28
Mf/mL
  12 Months | 20.70 [12.10 to 35.40] | 0.48 [0.07 to 3.10] | 1.30 [0.46 to 3.40] | 0.05 [0.01 to 0.42]
  24 Months: number analyzed (Participants) | 25 | 16 | 22 | 23
  24 Months | 8.10 [3.10 to 21.40] | 2.50 [0.57 to 10.60] | 2.00 [0.32 to 12.70] | 0.70 [0.12 to 4.20]

5. Secondary Outcome: Reduction in Circulating Filarial Antigen (CFA) Counts
Description: Reduction in circulating filarial antigen (CFA) counts (relative to baseline) at 12 & 24 months
Time Frame: Assessed at Baseline, 6, 12, & 24 months; 12 and 24 months reported
Population: Geometric mean of circulating filarial antigen ng/mL at 12 and 24 months
Measure: Geometric Mean (95% Confidence Interval); unit: ng/mL
Arm/Group | IA (Ivermectin + Albendazole) | MoxA (Moxidectin + Albendazole) | IDA (Ivermectin + Diethylcarbamazine + Albendazole) | MoxDA (Moxidectin + Diethylcarbamazine + Albendazole)
Number analyzed (Participants) | 25 | 19 | 28 | 28
ng/mL
  12 Months | 21.70 [13.60 to 34.60] | 12.50 [7.30 to 21.40] | 10.30 [6.60 to 16.20] | 7.80 [4.80 to 12.60]
  24 Months | 12.16 [7.53 to 19.65] | 6.38 [3.7 to 11.01] | 5.14 [3.16 to 8.69] | 4.76 [2.89 to 7.84]

6. Secondary Outcome: Inactivation of Adult Worm Nests in Male Participants Only
Description: Inactivation of adult worm nests as assessed by scrotal ultrasound at 6, 12, and 24 months after treatment in male participants only
Time Frame: 6, 12, & 24 months
Population: Participants with worm nest clearance (MALES ONLY)
Measure: Count of Participants; unit: Participants
Arm/Group | IA (Ivermectin + Albendazole) | MoxA (Moxidectin + Albendazole) | IDA (Ivermectin + Diethylcarbamazine + Albendazole) | MoxDA (Moxidectin + Diethylcarbamazine + Albendazole)
Number analyzed (Participants) | 25 | 19 | 28 | 26
Participants
  12 Months: number analyzed (Participants) | 16 | 11 | 13 | 14
  12 Months | 1 | 7 | 10 | 10
  24 Months: number analyzed (Participants) | 16 | 9 | 9 | 12
  24 Months | 4 | 8 | 7 | 12

7. Secondary Outcome: Frequency and Severity of AEs
Description: Frequency and severity of AEs during the first 7 days after treatment.
Time Frame: From baseline treatment to 7 days post-treatment
Population: Frequency of AEs
Measure: Count of Participants; unit: Participants
Arm/Group | IA (Ivermectin + Albendazole) | MoxA (Moxidectin + Albendazole) | IDA (Ivermectin + Diethylcarbamazine + Albendazole) | MoxDA (Moxidectin + Diethylcarbamazine + Albendazole)
Number analyzed (Participants) | 41 | 40 | 41 | 42
Participants | 22 | 24 | 18 | 15

8. Secondary Outcome: Plasma Levels of Drugs/Metabolites Post Treatment
Description: Noncompartmental pharmacokinetic analyses of DEC, ABZ, ABZSO, ABZSO2, IVM and Mox concentrations will be conducted using WinNonlin (Pharsight Corporation; Cary, North Carolina, USA). Drug plasma concentrations and computed pharmacokinetic parameters will be listed by subject and summarized by drug or metabolite (geometric mean with coefficient of variation, arithmetic mean with standard deviation, minimum, maximum, number of observations). Individual and geometric mean (by time) concentrations versus time will be plotted for each treatment group on both linear and natural logarithm scales.
Time Frame: Baseline, 2, 3, 4, 6, 12, 24, & 48 hours post-treatment
Population: Dose Normalized AUC (ng*hr/mL)
Measure: Mean (95% Confidence Interval); unit: ng*hr/mL
Arm/Group | IA (Ivermectin + Albendazole) | MoxA (Moxidectin + Albendazole) | IDA (Ivermectin + Diethylcarbamazine + Albendazole) | MoxDA (Moxidectin + Diethylcarbamazine + Albendazole)
Number analyzed (Participants) | 15 | 15 | 14 | 14
ng*hr/mL
  ALB | 116.2 [10 to 686.3] | 172.1 [8 to 648.7] | 124.2 [9.9 to 366.2] | 82.4 [12.9 to 386.6]
  ALB-OX | 3302.3 [1355.5 to 11146.8] | 4078.9 [897.4 to 5738.5] | 3512.5 [1264.8 to 9680.3] | 2595.8 [897.4 to 5738.5]
  ALB-ON | 187.3 [43.2 to 593.9] | 300.8 [89.2 to 775] | 217.1 [79.5 to 613.5] | 174 [89.4 to 466.2]
  DEC: number analyzed (Participants) | 0 | 0 | 14 | 14
  DEC |  |  | 21308.2 [11177.4 to 28869.3] | 19544.9 [12412.9 to 28740.7]
  IVM: number analyzed (Participants) | 15 | 0 | 14 | 0
  IVM | 1505.1 [606.5 to 3318.4] |  | 1690.9 [885.5 to 3222.2] |
  MOX: number analyzed (Participants) | 0 | 15 | 0 | 14
  MOX |  | 2530.8 [549.2 to 5933.8] |  | 2653.2 [993.5 to 7507.8]

ADVERSE EVENTS:
Time Frame: Active adverse event monitoring took place from treatment to 7 days post-treatment. Passive adverse event monitoring continued through 36-months.
Arm/Group | IA (Ivermectin + Albendazole) | MoxA (Moxidectin + Albendazole) | IDA (Ivermectin + Diethylcarbamazine + Albendazole) | MoxDA (Moxidectin + Diethylcarbamazine + Albendazole)
All-Cause Mortality (participants affected / at risk) | 0/41 | 2/40 | 2/41 | 0/42
Serious Adverse Events (participants affected / at risk) | 0/41 | 2/40 | 2/41 | 0/42
Other Adverse Events (participants affected / at risk) | 22/41 | 24/40 | 18/41 | 15/42
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | IA (Ivermectin + Albendazole) (N=41) | MoxA (Moxidectin + Albendazole) (N=40) | IDA (Ivermectin + Diethylcarbamazine + Albendazole) (N=41) | MoxDA (Moxidectin + Diethylcarbamazine + Albendazole) (N=42)
Death (General disorders) | 0 | 1 | 2 | 0 — Fatal SAE
Seizure (General disorders) | 0 | 1 | 0 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | IA (Ivermectin + Albendazole) (N=41) | MoxA (Moxidectin + Albendazole) (N=40) | IDA (Ivermectin + Diethylcarbamazine + Albendazole) (N=41) | MoxDA (Moxidectin + Diethylcarbamazine + Albendazole) (N=42)
Abdominal Pain (Gastrointestinal disorders) | 7 | 2 | 4 | 2
Cough (General disorders) | 2 | 0 | 0 | 2
Diarrhea (General disorders) | 5 | 3 | 3 | 4
Difficulty Breathing (General disorders) | 0 | 0 | 0 | 1
Dizziness, giddiness, or fainting (General disorders) | 5 | 1 | 1 | 4
Fatigue (General disorders) | 1 | 2 | 0 | 1
Headache (General disorders) | 9 | 4 | 3 | 5
Itching Skin (General disorders) | 2 | 7 | 0 | 2
Muscle or Joint Pain (General disorders) | 5 | 11 | 5 | 5
Nausea (General disorders) | 0 | 0 | 3 | 1
Swollen or Painful Nodules (General disorders) | 0 | 0 | 1 | 0
Testicular or Scrotal Pain (General disorders) | 0 | 0 | 3 | 3
Vomiting (General disorders) | 0 | 0 | 1 | 0
Other (General disorders) | 0 | 0 | 3 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-06-01): https://cdn.clinicaltrials.gov/large-docs/06/NCT04410406/Prot_SAP_000.pdf